CLINICAL TRIAL: NCT05758987
Title: Evaluation of Blended CBT for PTSD in Regular Care: A New Format of Computer-Assisted Trauma-Focused Cognitive Behavioral Therapy: A Randomized Controlled Non-inferiority Trial
Brief Title: Blended Treatment för PTSD: A New Format of Computer-Assisted Trauma-Focused Cognitive Behavioral Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Capio Group (Other); Stockholm University (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Sigrid Salomonsson, Principal investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-07130
Record Dates: First submitted 2023-02-15; First posted 2023-03-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: PTSD; CBT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: A randomized controlled non-inferiority trial evaluating if the new blended Tf-CBT is non inferior to the gold standard PTSD treatment Prolonged exposure. The trial is a multicenter study conducted at 3-6 sites. Participants are individually randomized in blocks of 2-4 at each site.
Who Masked: Outcomes Assessor
Masking Description: Assessor of secondary outcome CAPS will be masked to participant allocation at post and follow-up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended Trauma focused Cognitive Behavioral Therapy (B-Tf-CBT) (Experimental): B-Tf-CBT shares key features with Internet-based CBT (I-CBT) in that it is based on a digital support accessible to the patient. This digital support equips blended treatment with the same proposed advantages as I-CBT in terms of improving treatment accessibility, adherence, and reducing therapist-time. In addition, incorporating 6 biweekly face-to-face sessions to facilitate and augment delivery of more demanding components of TF-CBT such as memory exposure.
  Interventions: Behavioral: Blended Trauma focused Cognitive Behavioral Therapy (B-Tf-CBT)
- Prolonged exposure (Active Comparator): Gold standard Tf-CBT Prolonged exposure will constitute the control condition. Prolonged exposure will be delivered by trained therapists under supervision adhering to the evidence based manual delivered face-to-face over 9-15 weeks.
  Interventions: Behavioral: Prolonged exposure

INTERVENTIONS:
Behavioral: Blended Trauma focused Cognitive Behavioral Therapy (B-Tf-CBT) — A trauma-focused CBT where internet-based treatment is blended with face-to-face sessions with a therapist.
  Arms: Blended Trauma focused Cognitive Behavioral Therapy (B-Tf-CBT)
Behavioral: Prolonged exposure — A gold standard trauma-focused CBT delivered with face-to-face sessions with a therapist.
  Arms: Prolonged exposure

SUMMARY:
A Randomized Controlled Non-inferiority Trial testing if the new experimental Blended Trauma focused cognitive behavioral therapy (B-TF-CBT) for post traumatic stress disorder (PTSD), is non-inferior to gold standard control treatment Prolonged Exposure (PE).

Research question and hypothesis

Primary

1. Is bTF-CT non-inferior to prolonged exposure (PE) when delivered in routine clinical care in terms of PTSD symptoms on the PCL-5 post-treatment?

   Secondary:
2. Is bTF-CT non-inferior to prolonged exposure (PE) when delivered in routine clinical care in terms of PTSD symptoms on the PCL-5 at 6 and 12 months follow up?
3. Are there significant differences between bTF-CT and PE when delivered in routine clinical care in terms of depression, anxiety, insomnia, functionality, complex PTSD, other PTSD-measures and treatment satisfaction post-treatment and at 6 and 12 months follow up?

The study will be conducted at 3-6 outpatient clinics in Region Stockholm, Sweden.

DETAILED DESCRIPTION:
To study effects, the investigators aim to conduct a randomized controlled trial (RCT) comparing blended treatment to an evidence-based face-to-face TF-CBT protocol, Prolonged exposure.

Data will be collected concerning symptoms of PTSD with the PTSD Checklist for Diagnostic and Statistical Manual 5 (DSM-5; PCL-5) which will be the primary outcome measure. Further, symptoms of PTSD will be measured with Clinician-administered PTSD Scale for DSM-5 (CAPS-5), depression The PHQ-9, symptoms of anxiety with GAD-7 , quality of life with Work and social adjustment scale (WSAS), and sleep with the insomnia severity index (ISI). Outcome measures will be distributed before, during, after, as well as 12-months following treatment.

In accordance with CONSORT recommendations for non-inferiority trials, both intention-to-treat (ITT) and per-protocol (PP) analyses will be performed and reported for the primary non-inferiority comparisons. Secondary outcomes will be analyzed using ITT principles.

ITT population All randomized participants who completed the pre-treatment assessment and participated in the inclusion session.

PP population The PP population will include participants who have received at least 50% of the planned total treatment dose, defined across both digital modules and face-to-face sessions in the blended format.

Demographic variables Basic demographic variables (e.g., age, gender, education, trauma history, employment, and comorbid psychiatric disorders) will be collected at baseline.

Therapist competence and fidelity Therapist competence and adherence to PE and blended TF-CBT protocols will be assessed using structured fidelity checklists. A subset of recorded sessions will be rated by independent assessors.

Inter-rater reliability for CAPS-5 Interrater reliability will be assessed by having all CAPS raters independently score the same recorded role-play CAPS interview, with agreement evaluated using intraclass correlation coefficients (ICC), both between raters and relative to a predefined reference rating

Protocol deviations and adverse events Protocol deviations and adverse events (e.g., treatment interruptions, medication changes, unexpected events) will be documented and summarized descriptively.

Treatment dose and engagement Treatment engagement (e.g., number of sessions, digital module completion, total therapeutic time, and treatment duration) will be recorded to describe dose and support per-protocol analyses.

Concurrent treatments Participants will be asked about any concurrent psychological or pharmacological treatment at follow-up assessments.

To analyze the data, a non-inferiority analysis will be applied for the primary outcome variable. Step one in this analysis will be to determine what difference in mean scores on the PCL-5 between the two treatments is tolerated to conclude that the experimental intervention is non-inferior to the standard treatment (non-inferiority margin). Continuous outcomes will be analysed using linear mixed models, and non-inferiority will be assessed based on the 95% confidence interval for the estimated mean difference between treatments. Non-inferiority will be concluded if the lower bound of the confidence interval for the experimental treatment (bTF-CT) is above the predefined non-inferiority margin. If this criterion is met, the experimental treatment will be interpreted as non-inferior to the standard treatment (TF-CBT).

The non-inferiority margin was determined using procedures recommended in methodological guidelines for non-inferiority trials. One approach was based on preservation of a proportion of the established effect of the active control. Specifically, a pooled effect size of 1.0 for prolonged exposure therapy (PE) was identified from a published meta-analysis. In accordance with recommended practice, 50% of this effect was retained to define the non-inferiority margin, corresponding to a Cohen's d of 0.5. To adopt a more conservative approach and to ensure that the margin remained below the conventional threshold for a medium-sized effect, the non-inferiority margin was therefore set to Cohen's d = 0.4. Assuming a standard deviation of 15.98 on the PCL-5, based on post-treatment values from a comparable reference study, this corresponds to an absolute mean difference of approximately 7 points on the PCL-5. This value was therefore selected as the non-inferiority margin. As an additional check of clinical plausibility, the selected margin was compared with previously established estimates of the minimal important difference (MID) for the PCL-5, which have been reported to be approximately 9 points, indicating that the chosen margin was conservative.

Further, to estimate the required sample size, rigorous power calculations were carried out in collaboration with an expert in statistical analysis, applying a simulation-based approach using a 2-level linear mixed-effects model, using estimates from the reference TF-CBT, looking at six assessment points. Variance components that were incorporated into the analysis were random intercept, random slopes and residual variance. The power calculation showed that with 78 participants in each treatment group and a 20% dropout rate, 80% power is reached, given a non-inferiority margin of 7 points and α = 0.05.

An interim power analysis was also conducted by an external analyst, using model parameters from observed data in the power analysis, while also updating the number of assessment points to 16 and using α = 0.025. This resulted in 70 participants per group with power > 80%. To allow for per-protocol analysis, we will aim for 160 participants in total.

Continuous outcomes will be analyzed using linear mixed models (LMM) with an appropriate distribution family. Model checks for residuals and outliers will be performed using the R packages 'DHARMa' and 'performance' with default settings. If outliers are identified, this will be handled by using a robust LMM. Time in weeks will be treated as a continuous linear variable. The baseline measurement will be used as a covariate, modeled with a restricted cubic or natural spline. If time is found to be non-linear, it will also be modeled using splines. Confidence intervals will be generated using bootstrap. The mean difference between intervention groups (average treatment effect) will be estimated for the post-treatment measurement point using g-estimation. In the main analysis, treatment site will be added as a fixed effect covariate interacted with the treatment variable, and a therapist variable using a random slope only. This analysis will be conducted both using intent-to-treat (ITT) and per-protocol (PP). Missing data will be handled by multiple imputation with chained equations, imputing 20 datasets for analysis and pooling results. If there are differences in adherence between treatment groups for the PP analysis, a more robust method will be used, such as inverse probability of treatment weighting of instrumental variables(1). The investigators will also calculate effect sizes using Cohen's d based on pooled standard deviations.

Following regulatory recommendations (2), a baseline covariate-adjusted analysis will also be conducted and reported. This model will use the ANHECOVA approach, where all covariates interact with the treatment variable. Planned covariates that are added compared to the main analysis are: age, gender, education level, depression score, insomnia severity index score, work and social adjustment scale score, and trauma during childhood. Continuous baseline variables will be grand mean centered. Bootstrap will be used for confidence intervals. This analysis will only use ITT.

Sensitivity analyses will be conducted. One model will include only baseline, mid-treatment and post-treatment measurement points, since these are expected to have much lower attrition compared to weekly measurements. We will use a mixed model for repeated measurements (MMRM) with an unstructured covariance matrix. This model will also be fitted using both ITT and PP. The credibility and expectancy scale (CEQ), measured 2 weeks post-treatment start, will be used as a covariate in one model to evaluate potential effects of CEQ on the primary outcome. This model will also include the list of covariates specified in the previous paragraph.

Dichotomous variables that will be analyzed as outcomes: Remission rates will be calculated using a cut off of 31 on the PCL-5, across time in weeks; having a PTSD diagnosis according to CAPS-5 at time points pre, post, 6- and 12-months follow-up; and the proportion of patients who will show treatment response on the PCL-5, defined as a reduction of at least 10 points from baseline. All dichotomous outcomes will be analyzed using mixed model logistic regressions and comparisons between treatment groups will be reported as incident rate ratios and/or risk differences. Dichotomous data of remission will also be analyzed with survival analysis where time to remission is calculated and compared between groups.

1. Dodd M, Carpenter J, Thompson JA, et al. Assessing efficacy in non-inferiority trials with non-adherence to interventions: Are intention-to-treat and per-protocol analyses fit for purpose? Stat Med 2024; 43: 2314-2331. DOI: https://doi.org/10.1002/sim.10067.
2. Ye T, Shao J, Yi Y, et al. Toward Better Practice of Covariate Adjustment in Analyzing Randomized Clinical Trials. Journal of the American Statistical Association 2023; 118: 2370-2382. DOI: 10.1080/01621459.2022.2049278.

ELIGIBILITY:
Inclusion Criteria:

* PTSD according to Diagnostic and Statistical Manual of mental disorders 5 as primary problem
* ≥ 18 years
* Basic knowledge of speaking and writing Swedish
* No other psychological treatment at the same time
* No ongoing threats or violence
* If antidepressant medication, stable dose 6 weeks before starting treatment
* Have access to the internet and a computer
* Willingness/ability to participate after receiving information about what participation entails

Exclusion Criteria:

* Other diagnosis or problem is assessed as primary to PTSD
* Moderate to severe suicidal risk
* PTSD from childhood trauma that the person cannot remember

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
The Posttraumatic stress disorder checklist 5 (PCL-5) | Change from pre intervention to immediately post intervention
  Self rated PTSD-symptoms. Minimum value 0, maximum value 80, where higher values indicate more PTSD symptoms.
The Posttraumatic stress disorder checklist 5 (PCL-5) | Change from pre intervention to 6 months post intervention
  Self rated PTSD-symptoms. Minimum value 0, maximum value 80, where higher values indicate more PTSD symptoms.
The Posttraumatic stress disorder checklist 5 (PCL-5) | Change from pre intervention to 12 months post intervention
  Self rated PTSD-symptoms. Minimum value 0, maximum value 80, where higher values indicate more PTSD symptoms.

SECONDARY OUTCOMES:
Clinician-administered PTSD Scale for DSM-5 (CAPS-5) | 1 week post intervention
  * The traumatic event.
  * The 20 PTSD symptoms according to DSM-5.
  * The onset of PTSD symptoms.
  * Duration of PTSD symptoms.
  * The degree of subjective discomfort and mental strain due to PTSD symptoms.
  * The degree of impairment in social, professional and other functioning due to PTSD symptoms.
  * The degree of symptom improvement since the previous CAPS assessment.
  * Reliability/validity of the client's responses (i.e. whether the responses are truthful).
  * Overall severity of the PTSD symptoms.
  * CAPS-5 contains estimates of dissociative subtypes (depersonalization and derealization) that are new to DSM-V (i.e., not included in DSM-IV criteria for PTSD).
  A 0-4 scale is used for each of the 30 items: (0 = absence of symptoms, 1 = mild/subthreshold, 2 = moderate/threshold, 3= severe/markedly elevated, 4 = extreme/disabling)
Clinician-administered PTSD Scale for DSM-5 (CAPS-5) | 12 months post intervention
  * The traumatic event.
  * The 20 PTSD symptoms according to DSM-5.
  * The onset of PTSD symptoms.
  * Duration of PTSD symptoms.
  * The degree of subjective discomfort and mental strain due to PTSD symptoms.
  * The degree of impairment in social, professional and other functioning due to PTSD symptoms.
  * The degree of symptom improvement since the previous CAPS assessment.
  * Reliability/validity of the client's responses (i.e. whether the responses are truthful).
  * Overall severity of the PTSD symptoms.
  * CAPS-5 contains estimates of dissociative subtypes (depersonalization and derealization) that are new to DSM-V (i.e., not included in DSM-IV criteria for PTSD).
  A 0-4 scale is used for each of the 30 items: (0 = absence of symptoms, 1 = mild/subthreshold, 2 = moderate/threshold, 3= severe/markedly elevated, 4 = extreme/disabling)
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to immediately post intervention
  The PHQ-9 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 27. Higher scores indicating more symptoms. The first nine items in the PHQ-9 correspond to the nine criteria for depression in the DSM-IV. The tenth item is a simple function scale.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV. You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps for the first 9 items are scored from 0 to 3 and summed.
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to 6 months post intervention
  The PHQ-9 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 27. Higher scores indicating more symptoms. The first nine items in the PHQ-9 correspond to the nine criteria for depression in the DSM-IV. The tenth item is a simple function scale.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV. You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps for the first 9 items are scored from 0 to 3 and summed.
Patient Health Questionnaire (PHQ-9) | Change from pre intervention to 12 months post intervention
  The PHQ-9 is a brief self-rating scale for screening major depression according to DSMIV and measuring current symptom level of depression. Min 0 max 27. Higher scores indicating more symptoms. The first nine items in the PHQ-9 correspond to the nine criteria for depression in the DSM-IV. The tenth item is a simple function scale.
  The scale can be used as screening for the criteria for a depressive syndrome may be present according to DSM-IV. You can also use the sum score as a measure of the current level of symptoms to assess the depth of depression and follow a course over time. The scale steps for the first 9 items are scored from 0 to 3 and summed.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre intervention to immediately post intervention
  The GAD-7 is an instrument developed to help people who have anxiety symptoms that can be described as GAD. The test is only indicative and can never replace a doctor's visit and accurate diagnostics. The questions can be a help for the customer to identify any problems together with their doctor.
  If the client is already undergoing treatment for GAD, it may also be valuable to do a self-assessment from time to time to evaluate the effect of the treatment. A good opportunity can be in connection with and before a return visit to a doctor or psychologist or alternatively in connection with the renewal of a prescription. The customer can print out and take the test result to their doctor.
  The seven questions are scored from 0 (Not at all) to 3 (Daily) and summed. The total score is thus within the range 0-21.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre intervention to 6 months post intervention
  The GAD-7 is an instrument developed to help people who have anxiety symptoms that can be described as GAD. The test is only indicative and can never replace a doctor's visit and accurate diagnostics. The questions can be a help for the customer to identify any problems together with their doctor.
  If the client is already undergoing treatment for GAD, it may also be valuable to do a self-assessment from time to time to evaluate the effect of the treatment. A good opportunity can be in connection with and before a return visit to a doctor or psychologist or alternatively in connection with the renewal of a prescription. The customer can print out and take the test result to their doctor.
  The seven questions are scored from 0 (Not at all) to 3 (Daily) and summed. The total score is thus within the range 0-21.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre intervention to 12 months post intervention
  The GAD-7 is an instrument developed to help people who have anxiety symptoms that can be described as GAD. The test is only indicative and can never replace a doctor's visit and accurate diagnostics. The questions can be a help for the customer to identify any problems together with their doctor.
  If the client is already undergoing treatment for GAD, it may also be valuable to do a self-assessment from time to time to evaluate the effect of the treatment. A good opportunity can be in connection with and before a return visit to a doctor or psychologist or alternatively in connection with the renewal of a prescription. The customer can print out and take the test result to their doctor.
  The seven questions are scored from 0 (Not at all) to 3 (Daily) and summed. The total score is thus within the range 0-21.
Insomnia Severity Index (ISI) | Change from pre intervention to immediately post intervention
  A self-report questionnaire intended to measure insomnia. The purpose of the form is to quickly obtain a measure of the severity of sleep problems. The scale consists of 7 questions that evaluate falling asleep, sleep during the night, early awakening, the feeling of being rested, how sleep problems affect daily life and how the sleep pattern worries the individual. For each question, the participants must take a position on how they have experienced their sleeping habits in the past two weeks and then indicate the answers on a five-point Likert scale from 0 to 4, where 0 stands for "not at all" and 4 stands for "very much". The points are then added up. The total can be from 0 to 28 points. High scores indicate more severe sleep problems.
Insomnia Severity Index (ISI) | Change from pre intervention to 6 months post intervention
  A self-report questionnaire intended to measure insomnia. The purpose of the form is to quickly obtain a measure of the severity of sleep problems. The scale consists of 7 questions that evaluate falling asleep, sleep during the night, early awakening, the feeling of being rested, how sleep problems affect daily life and how the sleep pattern worries the individual. For each question, the participants must take a position on how they have experienced their sleeping habits in the past two weeks and then indicate the answers on a five-point Likert scale from 0 to 4, where 0 stands for "not at all" and 4 stands for "very much". The points are then added up. The total can be from 0 to 28 points. High scores indicate more severe sleep problems.
Insomnia Severity Index (ISI) | Change from pre intervention to 12 months post intervention
  A self-report questionnaire intended to measure insomnia. The purpose of the form is to quickly obtain a measure of the severity of sleep problems. The scale consists of 7 questions that evaluate falling asleep, sleep during the night, early awakening, the feeling of being rested, how sleep problems affect daily life and how the sleep pattern worries the individual. For each question, the participants must take a position on how they have experienced their sleeping habits in the past two weeks and then indicate the answers on a five-point Likert scale from 0 to 4, where 0 stands for "not at all" and 4 stands for "very much". The points are then added up. The total can be from 0 to 28 points. High scores indicate more severe sleep problems.
The Work and Social Adjustment Scale (WSAS) | Change from pre intervention to immediately post intervention
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better.
  The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
The Work and Social Adjustment Scale (WSAS) | Change from pre intervention to 6 months post intervention
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better.
  The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
The Work and Social Adjustment Scale (WSAS) | Change from pre intervention to 12 months post intervention
  The WSAS is a simple, reliable and valid measure of impaired functioning. It is a sensitive and useful outcome measure offering the potential for readily interpretable comparisons across studies and disorders. The maximum score of the WSAS is 40, lower scores are better.
  The 5 items are scored 0-8 ranging from Not at-all-Slightly-Definitely-Markedly-Very-severely
EUROQOL 5 dimensions (EQ5D) | Change from pre intervention to immediately post intervention
  The EQ-5D [1] is an instrument that consists of two parts and measures health-related quality of life, regardless of disease profile. The instrument measures the general state of health within five dimensions. Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. An EQ-5D value is also sometimes known as an 'index', 'score' or 'utility'.
EUROQOL 5 dimensions (EQ5D) | Change from pre intervention to 6 months post intervention
  The EQ-5D [1] is an instrument that consists of two parts and measures health-related quality of life, regardless of disease profile. The instrument measures the general state of health within five dimensions. Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. An EQ-5D value is also sometimes known as an 'index', 'score' or 'utility'.
EUROQOL 5 dimensions (EQ5D) | Change from pre intervention to 12 months post intervention
  The EQ-5D [1] is an instrument that consists of two parts and measures health-related quality of life, regardless of disease profile. The instrument measures the general state of health within five dimensions. Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. An EQ-5D value is also sometimes known as an 'index', 'score' or 'utility'.
Questions about work situation | Pre intervention
  Self constructed questions regarding work, employment and sick leave to evaluate in what degree the participant has worked the last 6 months
Questions about work situation | 6 months post intervention
  Self constructed questions regarding work, employment and sick leave to evaluate in what degree the participant has worked the last 6 months
Questions about work situation | 12 months post intervention
  Self constructed questions regarding work, employment and sick leave to evaluate in what degree the participant has worked the last 6 months
Registry data for the cost-effectiveness analysis | During the 12 month period post intervention
  * From the Center for Health Data: Variables on care consumption in primary care, inpatient care and outpatient care, including ambulance transports, medication prescription
  * From the National Board of Health and Welfare: Assistance decision Home help & help in the home.
  * From the Swedish Social Insurance Agency: Sick leave
Posttraumatic cognitions inventory (PTCI) | Pre intervention
  The Posttraumatic Cognitions Inventory measures negative PTSD-related cognitions about self, others and guilt. 36 items rated from 1 = Strongly disagree; 2 = Strongly Disagree; 3 = Disagree to some extent; 4 = Neutral; 5 = Agree to some extent; 6 = Agree to a large extent; 7 = Completely agree
Posttraumatic cognitions inventory (PTCI) | 6 weeks post intervention start
  The Posttraumatic Cognitions Inventory measures negative PTSD-related cognitions about self, others and guilt. 36 items rated from 1 = Strongly disagree; 2 = Strongly Disagree; 3 = Disagree to some extent; 4 = Neutral; 5 = Agree to some extent; 6 = Agree to a large extent; 7 = Completely agree
Posttraumatic cognitions inventory (PTCI) | immediately post intervention
  The Posttraumatic Cognitions Inventory measures negative PTSD-related cognitions about self, others and guilt. 36 items rated from 1 = Strongly disagree; 2 = Strongly Disagree; 3 = Disagree to some extent; 4 = Neutral; 5 = Agree to some extent; 6 = Agree to a large extent; 7 = Completely agree
Posttraumatic cognitions inventory (PTCI) | 6 months post intervention
  The Posttraumatic Cognitions Inventory measures negative PTSD-related cognitions about self, others and guilt. 36 items rated from 1 = Strongly disagree; 2 = Strongly Disagree; 3 = Disagree to some extent; 4 = Neutral; 5 = Agree to some extent; 6 = Agree to a large extent; 7 = Completely agree
Posttraumatic cognitions inventory (PTCI) | 12 months post intervention
  The Posttraumatic Cognitions Inventory measures negative PTSD-related cognitions about self, others and guilt. 36 items rated from 1 = Strongly disagree; 2 = Strongly Disagree; 3 = Disagree to some extent; 4 = Neutral; 5 = Agree to some extent; 6 = Agree to a large extent; 7 = Completely agree
The Response to Intrusions Questionnaire (RIQ) | Pre intervention
  A 19-item inventory that assesses the use of dysfunctional cognitive and behavioral strategies in response to intrusions of the trauma. Each item is self-rated from 0-3 and summarized. Lower scores indicating less intrusions.
The Response to Intrusions Questionnaire (RIQ) | 6 weeks post intervention start
  A 19-item inventory that assesses the use of dysfunctional cognitive and behavioral strategies in response to intrusions of the trauma. Each item is self-rated from 0-3 and summarized. Lower scores indicating less intrusions.
The Response to Intrusions Questionnaire (RIQ) | Immediately post intervention
  A 19-item inventory that assesses the use of dysfunctional cognitive and behavioral strategies in response to intrusions of the trauma. Each item is self-rated from 0-3 and summarized. Lower scores indicating less intrusions.
The Response to Intrusions Questionnaire (RIQ) | 6 months post intervention
  A 19-item inventory that assesses the use of dysfunctional cognitive and behavioral strategies in response to intrusions of the trauma. Each item is self-rated from 0-3 and summarized. Lower scores indicating less intrusions.
The Response to Intrusions Questionnaire (RIQ) | 12 months post intervention
  A 19-item inventory that assesses the use of dysfunctional cognitive and behavioral strategies in response to intrusions of the trauma. Each item is self-rated from 0-3 and summarized. Lower scores indicating less intrusions.
The internet intervention Patient Adherence Scale (iiPAS) | 6 weeks post intervention start
  A tool to measure adherence in internet-delivered behavioral interventions. 7 items rated from 0-4 and summarized. Lower scores indicating less adherence to treatment.
The internet intervention Patient Adherence Scale (iiPAS) | Immediately post intervention
  A tool to measure adherence in internet-delivered behavioral interventions. 7 items rated from 0-4 and summarized. Lower scores indicating less adherence to treatment.
Client Satisfaction Questionnaire (CSQ-8) | Immediately post intervention
  Self rated questionnaire to rate satisfaction with treatment. 8 items rated from 1-4 and summarized. Lower scores indicating less satisfaction. Scale ranging from 0-32
Negative Effects Questionnaire (NEQ) | Immediately post intervention
  self-rating form to measure negative effects of psychological treatment The NEQ consists of 20 statements that are answered on a 0-4 Likert scale. Furthermore, there is an open question to try to capture such negative effects that are not included in the self-report form, but which may be of theoretical or clinical relevance. In addition, the respondent is asked to answer whether the negative effects experienced were due to the treatment they underwent or other circumstances. The scale ranges from 0-80, higher scores indicate more negative effects. However the scale is more descriptive than designed to calculate negative effects
credibility/expectancy questionnaire | Two weeks post intervention start
  The Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) is the most widely used measure of treatment credibility and expectancy in psychotherapy research, and is a revision of the original scale developed by Borkovec and Nau (1972). This updated version contains 6 items rated on a 1-9 or a 0%-100% scale, depending upon the item. This revised scale, which was used in the present study, has been subjected to factor analysis, with results indicating that the items load onto two distinct factors of credibility and expectancy (Devilly & Borkovec, 2000). The first three items of the scale load onto the credibility factor and the final three items load onto the expectancy factor. Credibility scale ranges from 0-9 higher ratings indicate more credibility. Expectancy scale ranges from 0-100 higher ratings indicate more expectancy of treatment effect.
International Trauma Questionnaire | Pre intervention for participants included 2025
  The International Trauma Questionnaire (ITQ) assesses ICD-11 PTSD and Complex PTSD using 12 symptom items (six PTSD, six DSO), each rated on a 0-4 scale (0 = Not at all, 4 = Extremely). PTSD and DSO severity scores range from 0-24, with higher scores indicating greater symptom severity. The ITQ also includes three functional impairment items rated 0-4, used for diagnostic determination of probable PTSD/CPTSD according to ICD-11 criteria.
International Trauma Questionnaire | Immediately post intervention for participants included 2025
  The International Trauma Questionnaire (ITQ) assesses ICD-11 PTSD and Complex PTSD using 12 symptom items (six PTSD, six DSO), each rated on a 0-4 scale (0 = Not at all, 4 = Extremely). PTSD and DSO severity scores range from 0-24, with higher scores indicating greater symptom severity. The ITQ also includes three functional impairment items rated 0-4, used for diagnostic determination of probable PTSD/CPTSD according to ICD-11 criteria.
International Trauma Questionnaire | 6 months post intervention for participants included 2025
  The International Trauma Questionnaire (ITQ) assesses ICD-11 PTSD and Complex PTSD using 12 symptom items (six PTSD, six DSO), each rated on a 0-4 scale (0 = Not at all, 4 = Extremely). PTSD and DSO severity scores range from 0-24, with higher scores indicating greater symptom severity. The ITQ also includes three functional impairment items rated 0-4, used for diagnostic determination of probable PTSD/CPTSD according to ICD-11 criteria.
International Trauma Questionnaire | 12 months post intervention for participants included 2025
  The International Trauma Questionnaire (ITQ) assesses ICD-11 PTSD and Complex PTSD using 12 symptom items (six PTSD, six DSO), each rated on a 0-4 scale (0 = Not at all, 4 = Extremely). PTSD and DSO severity scores range from 0-24, with higher scores indicating greater symptom severity. The ITQ also includes three functional impairment items rated 0-4, used for diagnostic determination of probable PTSD/CPTSD according to ICD-11 criteria.
Autonomy, Flexibility, and Alliance Scale (study-specific measure) | Immediately post intervention for participants included 2025
  This study-specific self-report instrument assesses three process-related dimensions in blended CBT: Autonomy, Flexibility, and Therapeutic Alliance. The scale includes 8 items, each rated on a 7-point Likert scale (1 = "Do not agree at all" to 7 = "Completely agree"), with higher scores indicating greater levels of the respective construct.
  The measure consists of three subscales:
  Autonomy (3 items): perceived influence over treatment content and procedures.
  Flexibility (2 items): perceived ability to adapt timing, pace, and format of the treatment.
  Therapeutic Alliance (3 items): perceived emotional support, understanding, and shared goals with the therapist.
  Subscale scores are calculated as the mean or sum of their respective items; no total score is used.
Autonomy, Flexibility, and Alliance Scale (study-specific measure) | Immediately post intervention for participants included 2025
  This study-specific self-report measure assesses patients' perceived competence, learning, and ability to apply therapeutic skills following blended CBT for PTSD. The scale includes 9 items, each rated on a 7-point Likert scale (1 = "Do not agree at all" to 7 = "Completely agree"), with higher scores indicating greater perceived competence and learning.
  The measure captures patients' confidence in using treatment strategies, managing PTSD-related symptoms, approaching previously avoided situations, and engaging in valued activities. Scores are examined at the item or scale level; no predefined subscales or total score is used.
Autonomy, Flexibility, and Alliance Scale (study-specific measure) | 6 months post intervention for participants included 2025
  This study-specific self-report measure assesses patients' perceived competence, learning, and ability to apply therapeutic skills following blended CBT for PTSD. The scale includes 9 items, each rated on a 7-point Likert scale (1 = "Do not agree at all" to 7 = "Completely agree"), with higher scores indicating greater perceived competence and learning.
  The measure captures patients' confidence in using treatment strategies, managing PTSD-related symptoms, approaching previously avoided situations, and engaging in valued activities. Scores are examined at the item or scale level; no predefined subscales or total score is used.

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Salomonsson, PhD, Principal Investigator — Karolinska institute, clinical neuroscience
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No